CLINICAL TRIAL: NCT06785688
Title: The Effectiveness of Use an Energy Protector Aids for Improving the Lower Back Pain, Sports and Autonomic Nerve
Brief Title: Energy Protector Aids for Improving the Lower Back Pain, Sports and Autonomic Nerve
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Cheng-Hsin General Hospital (Other)
Responsible Party: Principal Investigator, Pei-Hung Liao, Assistant Professor, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 777(109-16)
Record Dates: First submitted 2023-05-22; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: the Effect of Infrared Rays Devices on Lower Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 experiment(50) (Active Comparator): Far-infrared Devices on Lower Back Pain keep 4times/week
  Interventions: Device: Protective gear irradiated by infrared rays
- 1 control (50) (Active Comparator): routine Nursing education after out patient department 60 people
  Interventions: Device: Protective gear irradiated by infrared rays

INTERVENTIONS:
Device: Protective gear irradiated by infrared rays — irradiated by infrared rays back brace

SUMMARY:
The purpose of this study is to explore the impact of Protective gear irradiated by infrared rays intervention on back pain, motor protection and autonomic nerves.

DETAILED DESCRIPTION:
Before and after the experimental control study design, each case, using the Chinese version of the simple pain scale and autonomic nerve measurement and exercise protection knowledge as a research tool, before and after the test (3 months after using the protective gear), collected Lower back pain level: changes in pain intensity and pain effects, and changes in autonomic and motor protection knowledge before and after testing. The research data uses SPSS for Windows 25.0 software package English version for data processing and analysis. The main statistics are Independent t test, Pair samples t test, Chi-square test and Odds ratio etc. It is expected that in the future, patients will be able to provide a safe and effective pain care and improve the quality of life, thereby reducing the recurrence rate of back pain and reducing the social cost of medical treatment

ELIGIBILITY:
inclusion criteria were: (1) individuals aged 20 to 80 with self-determined lower back pain who scored 3 points or higher on a brief pain scale; and (2) individuals accustomed to using far infrared devices for lower back pain.

excluded criteria were: Unconscious individuals were excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
back pain sereve & impact | contineous use back brace for 3 months
  check back pain degree

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei university of nursing and health science, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No